CLINICAL TRIAL: NCT01736995
Title: Family and Adolescent Motivational Incentives for Leveraging Youth
Acronym: FAMILY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA032723-01A1 (NIH)
Record Dates: First submitted 2012-11-05; First posted 2012-11-29 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Substance-Related Disorders
Keywords: Substance Abuse; Adolescents; Families; Functional Family Therapy; Cognitive Behavioral Therapy; Motivational Therapy; Contingency Management
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Motivational/Cog Beh Tx-Contingency Mgmt (Experimental): The group Motivational Enhancement Tx/Cognitive Behavioral Tx (MET/CBT) treatment is a peer-focused, multi-component intervention involving 2 initial individual motivational sessions followed by 12 group sessions that includes a functional analysis of behavior to identify antecedents and consequences of drug use and skills training for coping with cravings, enhancing assertive communication, drug refusal, managing negative moods, problem-solving, decision-making, and relapse prevention. The additional inclusion of contingency management (CM) methods will provide immediate, tangible reinforcers as a consequence delivered contingently upon evidence of abstinence from substance use or other desirable behavior.
  Interventions: Behavioral: Contingency Management
- Functional Family Tx- Contingency Mgmt (Experimental): Functional Family Therapy (FFT) is a brief treatment for youth with problem behaviors, including substance abuse that consists of 12 to 14 weekly family sessions. The FFT treatment is applied in five distinct phases: Engagement, Motivation, Relational Assessment, Behavior Change, and Generalization and each phase has specific goals, techniques, and therapist skills. The additional inclusion of contingency management (CM) methods will provide immediate, tangible reinforcers to the family as a consequence delivered contingently upon evidence of abstinence from substance use or other desirable behavior.
  Interventions: Behavioral: Functional Family Therapy; Behavioral: Contingency Management
- Motivational/Cog Beh Tx (Experimental): The group Motivational Enhancement Tx/Cognitive Behavioral Tx (MET/CBT) treatment is a peer-focused, multi-component intervention involving 2 initial individual motivational sessions followed by 12 group sessions that includes a functional analysis of behavior to identify antecedents and consequences of drug use and skills training for coping with cravings, enhancing assertive communication, drug refusal, managing negative moods, problem-solving, decision-making, and relapse prevention.
  Interventions: Behavioral: Motivational Enhancement Tx/Cognitive Behavioral Tx
- Functional Family Tx (Experimental): Functional Family Therapy (FFT) is a brief treatment for youth with problem behaviors, including substance abuse that consists of 12 to 14 weekly family sessions. The FFT treatment is applied in five distinct phases: Engagement, Motivation, Relational Assessment, Behavior Change, and Generalization and each phase has specific goals, techniques, and therapist skills.
  Interventions: Behavioral: Functional Family Therapy

INTERVENTIONS:
Behavioral: Functional Family Therapy
  Other Names: FFT
  Arms: Functional Family Tx; Functional Family Tx- Contingency Mgmt
Behavioral: Motivational Enhancement Tx/Cognitive Behavioral Tx
  Other Names: MET/CBT
  Arms: Motivational/Cog Beh Tx
Behavioral: Contingency Management
  Other Names: CM
  Arms: Functional Family Tx- Contingency Mgmt; Motivational/Cog Beh Tx-Contingency Mgmt

SUMMARY:
Research has provided support for the efficacy of cognitive-behavioral and family interventions for adolescent substance use disorders (SUD), HIV-risk behaviors, and related problems. Despite support for these interventions, substantial heterogeneity in treatment outcomes and high relapse rates has been consistently found across studies. Such variability highlights the need for innovative strategies to broaden the impact and strengthen the durability of effects of adolescent substance abuse treatments. Over the past two decades, research has shown the positive effects of contingency management (CM) methods on reductions in substance use and other problem behaviors. When combined with evidence-based practices, emerging research suggests that CM integration may also be effective for adolescent substance abusers. The proposed Stage II efficacy trial examines the integration of CM with two empirically-supported interventions: group MET/CBT and FFT. By comparing two intervention modalities (group vs. family, the study provides a unique opportunity to examine the robustness of the effects of CM across established adolescent treatments, and to compare change mechanisms that may account for treatment outcomes. In the proposed research, substance abusing adolescents (n = 160) will be randomly assigned either to FFT or group MET/CBT. Random assignment will also be used to determine whether or not youth will receive a CM condition that provides incentives for abstinence (i.e., clean urine screens) and treatment participation. The primary aim of the study is to examine the efficacy of an integrated CM intervention for the two evidence-based treatments for adolescents, MET/CBT and FFT, compared to these treatments without CM on drug abuse abstinence (a) during treatment (i.e., speed of effects) and (b) at post-treatment follow-up assessments (i.e., durability of effects). A second aim of the study is to evaluate the effects of CM on hypothesized mediators of the intervention effects in the MET/CBT and the FFT conditions. The investigators anticipate that the CM conditions, compared to the nonCM conditions, are more likely to accelerate the adolescent's motivation (1) to achieve abstinence, to attend and participate in treatment, and to complete homework assignments. The investigators will also examine the effects of the interventions on HIV-risk behaviors and expect that CM will demonstrate the largest reductions in HIV-risk behaviors compared to the nonCM conditions.

DETAILED DESCRIPTION:
Research has provided support for the efficacy of cognitive-behavioral and family interventions for adolescent substance use disorders (SUD), HIV-risk behaviors, and related problems. Despite support for these interventions, substantial heterogeneity in treatment outcomes and high relapse rates have been consistently found across studies. Such variability highlights the need for innovative strategies to broaden the impact and strengthen the durability of effects of adolescent substance abuse treatments. Over the past two decades, research has demonstrated the positive effects of contingency management (CM) methods on reductions in substance use and other problem behaviors such as HIV-risk, primarily with adults. CM has been shown to improve outcomes when combined with evidence-based practices and research is emerging to suggest that such integrations may also be effective for adolescent substance abusers. The proposed Stage II efficacy trial examines the integration of CM with two empirically-supported interventions: group MET/CBT and FFT. By comparing two intervention modalities (group vs. family, the study provides a unique opportunity to examine the robustness of the effects of CM across established adolescent treatments, and to compare change mechanisms that may account for treatment outcomes. In the proposed research, substance abusing adolescents (n = 160) will be randomly assigned either to FFT or group MET/CBT. Random assignment will also be used to determine whether or not youth will receive a CM condition that provides incentives for abstinence (i.e., clean urine screens) and treatment participation. Thus, participants will receive one of four intervention conditions, two with an integrated CM intervention (MET/CBT-CM, FFT-CM) and two without CM (MET/CBT, FFT). The study will employ a 2 (Incentives: CM, nonCM) x 2 (Modality: MET/CBT, FFT) x 5 (Time: Baseline, 2-, 4-, 8-, and 12-months post-randomization) factorial design. The primary aim of the study is to examine the efficacy of an integrated CM intervention for the two evidence-based treatments for adolescents, MET/CBT and FFT, compared to these treatments without CM on drug abuse abstinence (a) during treatment (i.e., speed of effects) and (b) at post-treatment follow-up assessments (i.e., durability of effects). A second aim of the study is to evaluate the effects of CM on hypothesized mediators of the intervention effects in the MET/CBT and the FFT conditions. The investigators anticipate that the CM conditions, compared to the nonCM conditions, are more likely to accelerate the adolescent's motivation (1) to achieve abstinence, to attend and participate in treatment, and to complete homework assignments. Exploratory analyses will examine differences between modalities (MET/CBT vs FFT) on the presumed mediators. The investigators expect that MET/CBT will produce greater improvements in adolescents' drug avoidance self-efficacy and FFT will produce greater improvements in family relationships. The investigators will also examine the effects of the interventions on HIV-risk behaviors and expect that CM will demonstrate the largest reductions in HIV-risk behaviors compared to the nonCM conditions.

The study addresses the question of whether adding a Contingency Management (CM) approach, in which adolescents are provided with a monetary incentive for providing clean urine, enhances the efficacy of two research-proven interventions for adolescent substance use. Specifically, the investigators compare if Functional Family Therapy (FFT) and Motivational Enhancement/Cognitive Behavioral Therapy (MET/CBT) combined with CM are better than either intervention alone. The investigators also explore the extent to which the addition of CM increases the speed with which adolescents achieve abstinence as well as the durability of these effects over time. The inclusion of two distinct forms of therapy also permits the investigation of how the interventions achieve their effects on adolescent drug use (e.g., improvements in family functioning in FFT vs. improvements in drug avoidance and self-efficacy skills in MET/CBT).

Specific Aim 1: To evaluate the efficacy of CM versus nonCM conditions delivered in the context of either group (MET/CBT) or family (FFT) treatments for substance abusing adolescents. The investigators will use two substance use dependent variables. The first variable assesses the presence or absence of illegal substances in urine samples collected weekly beginning at baseline and continuing during the 12-14 weeks of scheduled treatment. Urine samples will be collected at all post-randomization assessments. Although most of the adolescents are polydrug users, marijuana is the primary drug of abuse. The investigators anticipate that once weekly urine screens will be able to detect recent marijuana use. The Time Line Follow-back (TLFB) will be used to provide weekly estimates of drug use abstinence for a period from 3 months before to 12 months after randomization. Specifically, the investigators predict that the CM versus the nonCM conditions will produce a significant main effect increase in the number of weeks of drug use abstinence during the treatment phase (i.e., months 1-4; Hypothesis 1a) and during the post treatment period (i.e., 4-12 months; Hypothesis 1b).

Specific Aim 2: To evaluate the efficacy of CM versus nonCM on secondary behavioral outcomes. Specifically, The investigators predict that CM versus the nonCM conditions will be associated with significantly lower levels of sexually risky behaviors (Hypothesis 2a) and conduct problems (Hypothesis 2b) over time.

Specific Aim 3: To evaluate the effects of CM on hypothesized mediators of the MET/CBT and the FFT intervention effects. The investigators anticipate that the CM conditions are more likely than the nonCM conditions to accelerate the adolescent's motivation (1) to achieve abstinence, (2) to attend and participate in treatment, (3) to complete homework assignments. The SOCRATES scale will assess their motivation to achieve abstinence. Specifically, the investigators predict that youth receiving the CM versus nonCM will show higher rates of motivation for change at the 2-month assessment (Hypothesis 3a) and higher rates of treatment attendance and homework compliance (as measured by weekly therapist reports) over the course of treatment (Hypothesis 3b).

Exploratory Aims: The investigators will conduct exploratory analyses to examine if the number of continuous weeks of abstinence during treatment, adolescent's motivation to achieve abstinence, attendance, and homework compliance will mediate abstinence following treatment. Additional analyses will examine differences between modalities (MET/CBT vs FFT) on the presumed mediators: MET/CBT will produce greater improvements in adolescent's drug avoidance self-efficacy and FFT will produce greater improvements in family relationships (as measured by the FES). Improvements in drug avoidance self-efficacy and family relationships will mediate improvements in MET/CBT and FFT, respectively. The investigators will also explore potential differences within modality to determine if adding CM enhances the effects of each modalities impact on the presumed mediators of outcome. The results of these analyses will help determine if there is sufficient merit to warrant additional research into mechanisms of action within each modality. Finally, the investigators will conduct an informal cost-effectiveness analysis to derive preliminary estimates of the relative costs of each treatment modality, particularly with respect to treatment engagement/attendance and youth outplacement to restricted settings.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 17 years of age
* Meets DSM-IV diagnostic criteria for substance abuse or dependence
* Living at home with the participating parent
* Sufficient residential stability to permit probable contact at follow- up(e.g., not homeless at time of intake)

Exclusion Criteria:

* Evidence of psychotic or organic state of sufficient severity to interfere with the understanding of study instruments and procedures
* Deemed dangerous to self or others at intake
* Services other than outpatient treatment are required for the youth (e.g., inpatient, detoxification)
* Marijuana use is reported as being less than 13% of the previous 90 days

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Urine Assays - NIDA 12 Test Panel | Up to 12-months after randomization
  The NIDA 12 Test Panel is a card device with 12 finger-like prongs, dipped in a urine sample to screen for the presence or absence of illegal substances including AMP (amphetamine), BAR (barbiturates), BZO (benzodiazepines), COC (cocaine), M-AMP/MDMA (methamphetamine, ice, speed, ecstasy), MTD (methadone), MOR (morphine), OXY (Oxycodone), PCP, PPX (Propoxyphene), OPI (Opiates), THC (marijuana). Alcohol use will be measured using Saliva Screens (Alco-Screen 02), a simple, non-invasive, one-step test that provides results in four minutes and detects alcohol levels of .02 or greater.

SECONDARY OUTCOMES:
Timeline Followback semi-structured interview (TLFB) | Up to 12-months after randomization
  The TLFB will be used to determine the percent days of substance use (primary measure), excluding tobacco, as well as abstinence days and binge drinking days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Robbins, Ph.D., Principal Investigator — Oregon Research Institute; Functional Family Therapy, Inc.
Locations (1):
- Oregon Research Institute Center for Family and Adolescent Research, Albuquerque, New Mexico, United States